CLINICAL TRIAL: NCT04421976
Title: Driving Pressure for Early Postoperative Redistribution of Pulmonary Ventilation in Neurosurgery : A Prospective Randomized Controlled Trial
Brief Title: Driving Pressure in Neurosurgery
Acronym: DPNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Wei Zhang, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DP-Neurosurgery
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Neurosurgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional PEEP (Placebo Comparator): PEEP = 5 cmH2O
  Interventions: Procedure: PEEP
- Driving pressure (DP) guided-PEEP (Experimental): PEEP is increased from 2 to 10 cm H2O incrementally. Each PEEP level is maintained for 10 respiratory cycles, with DP in the last cycle recorded. Then the PEEP level producing the lowest DP will be identified and maintained intraoperatively.
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: PEEP — Driving pressure (DP) is calculated as "plateau pressure - PEEP". 10min after position adjustment, PEEP is increased from 2 to 10 cm H2O incrementally. Each PEEP level is maintained for 10 respiratory cycles, with DP in the last cycle recorded. Then the PEEP level producing the lowest DP will be identified and maintained intraoperatively.

SUMMARY:
The effect of driving pressure (DP)-guided positive end expiratory pressure (PEEP) on early postoperative pulmonary ventilation is to be determined for patients undergoing neurosurgery. Patients are recruited to receive volume controlled ventilation with either a fixed PEEP (5cmH2O) or DP titrated PEEP. Early postoperative regional distribution of lung ventilation, expressed as global inhomogeneity (GI) is evaluated by electrical impedance tomography (EIT), a noninvasive, radiation free modality. Center of ventilation (COV) by EIT, as well as the lung ultrasonography（LUS), perioperative ventilatory parameters, arterial oxygenation index (PaO2/FiO2) , serum indicators and postoperative pulmonary complications are secondary outcome variables.

DETAILED DESCRIPTION:
After screened for preoperative risk factors, 44 patients undergoing elective neurosurgery and planned to be extubated in the operating room are randomly assigned to two groups: (1) PEEP = 5cmH2O; (2) driving pressure (DP)-guided PEEP. The ventilation protocol consists of volume-controlled mechanical ventilation (Datex Ohmeda S/5 Advance; General Electric Company Healthcare, Helsinki, Finland) at a tidal volume (VT) of 8 ml/kg predicted body weight (PBW), fresh gas of 2 litre /min, inspiratory to expiratory ratio of 1:2, and a respiratory rate adjusted to normocapnia (arterial carbon dioxide partial pressure between 35 and 45 mmHg). For group 2, trial for the lowest DP was started 10 min after position adjustment by increasing PEEP from 2 to 10 cm H2O incrementally. DP was calculated as "plateau pressure - PEEP". Each PEEP level was maintained for 10 respiratory cycles, with DP in the last cycle recorded. Then the PEEP level producing the lowest DP was identified and maintained intraoperatively. A plateau pressure of no more than 30 cmH2O is targeted in each group. Early postoperative distribution of regional ventilation global inhomogeneity (GI) is the primary endpoint evaluated by EIT (electrical impedance tomography), which was performed by a trained technician who is blinded to randomization. Center of ventilation (COV) by EIT, lung ultrasonography（LUS) , and arterial blood gas are evaluated, with inflammatory and oxidative mediators tested from venous sample. Brain relaxation will be scored by the neurosurgeon. Postoperative pulmonary complications within 3 days are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent has been obtained
* Elective neurosurgery
* Expected ventilation duration > 2 hours
* Scheduled to be extubated in the operation
* American Society of Anesthesiologists (ASA) physical status >2

Exclusion Criteria:

* Mechanical ventilation of > 1 hour within the last 2 weeks before surgery
* Dysphagia resulting from preoperative cranial nerve damage
* Body mass index ≥ 35 kg/m2
* Acute respiratory failure (pneumonia, acute lung injury or acute respiratory distress syndrome)
* Emergency surgery
* Severe cardiac disease
* Progressive neuromuscular illness
* Pregnancy
* Refusal to participate
* Contradicted to EIT scan or lung ultrasound scan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-21 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
early postoperative overall spatial distribution of pulmonary ventilation | immediately after extubation
  global inhomogeneity index (GI): overall degree of spatial heterogeneity of ventilation. GI is measured by electrical impedance tomography (EIT). A smaller GI index represents a more homogeneous distribution, and a larger GI index indicates a more inhomogeneous ventilation.

OTHER OUTCOMES:
Melbourne Group Scale version 2 (MGS-2) | within the first 3 days after surgery
  Melbourne Group Scale version 2 (MGS-2): Temperature >38°C; White cell count >11.2 or use of respiratory antibiotics; Physician diagnosis of pneumonia or chest infection; Chest X-ray findings of atelectasis/consolidation; Production of purulent (yellow/green) sputum different from preoperative sputum; Positive results upon sputum microbiological analysis; oxygen saturation by pulse oximetry (SpO2)<90% in ambient air; Re-admission to or prolonged stay (>36 h) in the intensive care unit/high dependency unit for respiratory problems. A postoperative pulmonary complication (PPC) was diagnosed if 4 or more of the 8 factors were present.

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, MD,PHD, Study Director — Beijing Tiantan Hospital affiliated with Capital Medical University
Locations (1):
- Department of Anesthesiology,Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu F, Zhang W, Zhao Z, Xu X, Jian M, Han R. Effect of driving pressure on early postoperative lung gas distribution in supratentorial craniotomy: a randomized controlled trial. BMC Anesthesiol. 2023 May 22;23(1):176. doi: 10.1186/s12871-023-02144-7. PMID 37217882